CLINICAL TRIAL: NCT02287103
Title: Effect of Eating vs Skipping Breakfast on Postprandial Hyperglycemia After Subsequent Isocaloric Lunch and Dinner in Type 2 Diabetic Patients
Brief Title: Eating vs Skipping Breakfast on Postprandial Hyperglycemia After Lunch and Dinner in T2D
Acronym: SkippB-T2D
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Daniela Jakubowicz, Dr, Tel Aviv University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0160-14-WOMC
Record Dates: First submitted 2014-11-02; First posted 2014-11-10 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Breakfast
Keywords: Skipping Breakfast
MeSH Terms: conditions — Intermittent Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Skipping Breakfast (NoB) (Experimental): The patients in No B will omit the breakfast and will continue the overnight fast until lunch. Will eat only lunch and dinner. In YesB will eat all three meals
  Interventions: Other: Skipping Breakfast
- Eating Breakfast (YesB): (Active Comparator): The patients in YesB will eat all three mealswill consume three meals: breakfast, lunch and dinner
  Interventions: Other: Eating Breakfast

INTERVENTIONS:
Other: Skipping Breakfast — NoB: The patients will omit the breakfast, will continue the overnight fast until lunch, then will eat only lunch and dinner.
  Other Names: omitting breakfast
  Arms: Skipping Breakfast (NoB)
Other: Eating Breakfast — YesB: will eat all three meals
  Arms: Eating Breakfast (YesB):

SUMMARY:
Background: Skipping breakfast and/or overeating at evening, has been associated in type 2 diabetic (T2D) individuals, with higher BMI, visceral adiposity, hyperlipidemia, increased overall postprandial glycemia (PPHG) and higher HbA1c. The absence of breakfast is also associated with increased plasma free fatty acids (FFA) along the morning until lunch. High plasma FFA in turn are triggering factor of insulin resistance, by inhibiting insulin mediated glucose uptake in obese and T2D subjects The investigators therefore hypothesize that compared to eating breakfast the prolonged overnight fasting caused by the breakfast omission will result in increased postprandial glycemic response after subsequent isocaloric lunch and dinner in T2D individuals.

Objectives: With this aim will study T2D patients in randomized crossover design to consume in two separate days, either 3 standard isocaloric meals: Yes Breakfast condition (YesB) or omit breakfast: no breakfast condition (NoB) and consume only lunch and dinner with the same caloric content.

Methods and Study Design: The YesB intervention will consist on three identical meals coating 700 Kcal each: breakfast at 8:00, lunch at 13:00 and dinner at 19:00. The NoB intervention the breakfast will be omitted and the subject continue fasting until lunch. Then the participants will consume identical 700 kcal Lunch at 13:00 and 700 Kcal dinners at 19:00. The investigators will assess plasma glucose, insulin, C-peptide, GLP-1 and FFA with blood samples collected every 30 min up to 180 min after breakfast, lunch and dinner and at the same time point the blood samples will be collected after 8:00 when the breakfast will be omitted.

Expected results: The investigators expect that compared to NoB condition, in the YesB condition the postprandial response after lunch and dinner will be reduced for glucose and for FFA, while plasma insulin, C-peptide and GLP-1 postprandial response after lunch and dinner will be enhanced

DETAILED DESCRIPTION:
Background or Rationale Studies analyzing the postprandial glycemic response have shown that glucose tolerance display a clear diurnal variation with a progressive decline in carbohydrate tolerance toward the evening hours with more prolonged and higher postprandial glycemic response in the evening than in the morning.

Meal timing patterns, on the other hand, exerts strong entraining influence on clock gene regulation of hormones and enzymes i.e. insulin, GLP-1, involved in glucose metabolism and postprandial glycemia disrupting the diurnal variation of postprandial glycemia (PPG). It suggests the extent of post-prandial rise in plasma glucose depends not only upon the quantity and nature of food ingested, and on the clock gene regulated circadian hormonal rhythms, it also depends upon the metabolic state immediately prior to eating. Indeed, meal schedule non-aligned with the clock gene circadian rhythms, such as skipping breakfast and/or overeating at evening, has been associated, in T2D individuals, with higher BMI, visceral adiposity, hyperlipidemia, higher HbA1c and increased PPG despite same caloric intake. The absence of breakfast has been associated in obese and T2D subjects with increased plasma levels of free fatty acids (FFA) along the morning until the lunch, Chronic and acute increase of FFA plasma levels, has been reported as triggering factor of insulin resistance, by inhibition of insulin mediated stimulated glucose uptake and/or phosphorylation which develops 3-4 hours after raising of plasma FFA and by inhibition of glycogen synthase, the rate limiting enzyme of glycogen synthesis, which develops 4-6 hours after the rise of FFA. However the effect of eating vs skipping breakfast on postprandial glucose response after identical lunch and dinner has not been explored. It is therefore important to explore the influence of eating versus skipping breakfast on postprandial glucose, after lunch and dinner in T2D individuals. Concomitantly the investigators will assess after lunch and dinner plasma insulin, GLP-1 and FFA response after lunch and dinner in T2D individuals.

Expected results: The investigators expect that compared skipping breakfast condition, the eating breakfast condition will reduce postprandial plasma glucose and FFA response after lunch and dinner, while plasma insulin, C-peptide and GLP-1 after lunch and dinner will be enhanced Relevance of the study: If our hypothesis is confirmed it may be may be of practical benefit to people with Type 2 diabetes, a condition in which the reduction of PPHG at lunch and at dinner may result in improved HbA1c and might be also preventive of the risk for CVD Objectives: With this aim will study T2D patients in randomized crossover design to consume in two separate days, either 3 standard isocaloric meals: Yes Breakfast condition (YesB) or omit breakfast: no breakfast condition (NoB) and consume only lunch and dinner with the same caloric content.

Methods and Study Design: The YesB intervention will consist on three identical meals coating 700 Kcal each: breakfast at 8:00, lunch at 13:00 and dinner at 19:00. The NoB intervention the breakfast will be omitted and the subject continue fasting until lunch. Then the participants will consume identical 700 kcal Lunch at 13:00 and 700 Kcal dinners at 19:00. The investigators will assess plasma glucose, insulin, C-peptide, GLP-1 and FFA with blood samples collected every 30 min up to 180 min after breakfast, lunch and dinner and at the same time point the blood samples will be collected after 8:00 when the breakfast will be omitted.

ELIGIBILITY:
Inclusion Criteria:

* T2D since < 10 yrs, with HbA1c > 7 % and BMI: 26-34 kg/m2.
* Only naïve or treated with oral antidiabetic drugs and with anti-hypertensive and lipid-lowering medication will be included.
* Those treated with insulin or GLP-1 analogs or having major liver, heart or kidney illnesses will be excluded.

Exclusion Criteria:

1. Type 1 DM, secondary DM, gestational DM
2. Patients using insulin, TZDs
3. Patients using corticosteroid, herb medication or other medications affecting glucose tolerance
4. Renal dysfunction (Cr > 1.5mg/dL)
5. Hepatic dysfunction (LFT > x 3UNL)
6. Anemia (Hg > 10g/dL)
7. Ischemic heart disease, congestive heart failure
8. Severe diabetic complication (CRF, CVA, PDR, gastroparesis)
9. Infectious disease
10. Malignancy
11. Pregnant women

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-04; Primary Completion 2015-09 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Measure of plasma glucose | 5 weeks
  Postprandial glycemia

SECONDARY OUTCOMES:
Measure of plasma Insulin | 5 weeks
Measure of plasma GLP-1 | 5 weeks
Measure of free fatty acids (FFA) | 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Jakubowicz, MD, Principal Investigator — Diabetes Unit E. Wolfson Medical center Holon, Tel Aviv Israe
Locations (1):
- Diabetes Unit E. Wolfson Medical center, Holon, Tel Aviv, Israel

REFERENCES:
- [Derived] Allaf M, Elghazaly H, Mohamed OG, Fareen MFK, Zaman S, Salmasi AM, Tsilidis K, Dehghan A. Intermittent fasting for the prevention of cardiovascular disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013496. doi: 10.1002/14651858.CD013496.pub2. PMID 33512717